CLINICAL TRIAL: NCT02404389
Title: A Randomized, Vehicle Controlled, Active Comparator, Parallel Group Study to Evaluate Safety, Tolerability and Preliminary Efficacy of Topical LFX453 Formulations in Patients With Actinic Keratosis
Brief Title: Safety, Tolerability, and Efficacy Study of LFX453 in Actinic Keratosis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLFX453X2201
Record Dates: First submitted 2015-01-23; First posted 2015-03-31 (Estimated); Results first posted 2018-03-19 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2019-03

CONDITIONS: Actinic Keratosis
Keywords: Actinic keratosis, patients, topical, lesion count, clearance rate
MeSH Terms: conditions — Keratosis, Actinic | interventions — Therapies, Investigational

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- LFX453 0.1% NMC (Experimental): LFX453 0.1% nanomedicinal cream (NMC) Twice daily applications
  Interventions: Drug: Investigational Treatment
- LFX453 0.15% LCC (Experimental): LFX453 0.15% liquid crystal cream (LCC) Twice daily applications
  Interventions: Drug: Investigational Treatment
- Vehicle to NMC (Placebo Comparator): Vehicle to nanomedicinal cream (NMC) Twice daily applications
  Interventions: Drug: Investigational Treatment
- Vehicle to LCC (Placebo Comparator): Vehicle to liquid crystal cream (LCC) Twice daily applications
  Interventions: Drug: Investigational Treatment
- Aldara (Active Comparator): Aldara cream 3 applications per week
  Interventions: Drug: Active comparator

INTERVENTIONS:
Drug: Investigational Treatment — Topical application for two treatment cycles with twice daily applications, separated by a 4 week treatment pause and followed by 8 week treatment free follow-up.
  Arms: LFX453 0.1% NMC; LFX453 0.15% LCC; Vehicle to LCC; Vehicle to NMC
Drug: Active comparator — Topical treatment with Aldara 3 times per week. The group will be open-label, but however blinded to the efficacy assessor, and followed by 8 week treatment free follow-up.
  Arms: Aldara

SUMMARY:
This is a randomized, vehicle controlled, active comparator, parallel group, study with a total duration of 24 weeks including screening and follow-up. Study drug is applied topically for 2 cycles of 4 week treatment, separated by 4 weeks off-treatment. Assessors of study endpoints are blinded to treatment allocation.

ELIGIBILITY:
Key Inclusion Criteria:

* Male patients, and female patients of non-childbearing potential, age ≥ 18 to ≤ 75 years (at the time of the screening visit), and in general good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening
* Patients with at least five clinically typical, visible or palpable non-hyperkeratotic AK lesions within a contiguous area of 25 cm2, or within 2 areas for a maximum total of 25cm2, on the face (at least 2 cm from the periocular areas, lips, nares and ears) and/or balding scalp
* Presence of at least one additional visible or palpable non hyperkeratotic AK lesion outside of the selected area amenable to the collection of a skin biopsy, and located at least at 2 cm from the limits of the area to receive treatment
* Male patients had to agree to use adequate contraception for the duration of the study.

Key Exclusion Criteria:

* Known hypersensitivity to any constituents of the study drugs (including local anesthetics if consenting to biopsies) or known allergies to imiquimod or to drugs of similar chemical classes or history of serious allergic reaction.
* Presence of atopic dermatitis, eczema, psoriasis, rosacea or other possible confounding skin conditions on face or balding scalp even outside of the treatment area.
* Invasive tumors within the treatment area, e.g., merkel cell carcinoma, melanoma, squamous cell carcinoma (SCC), basal cell carcinoma, the latter being accepted if completely surgically removed.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant.
* History of hypertrophic scarring.
* Concurrent disease that suppresses the immune system.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-03-05 (Actual); Primary Completion 2016-01-27 (Actual); Study Completion 2016-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- Novartis Investigative Site, Vienna, Austria
- Novartis Investigative Site, Copenhagen NV, Denmark
- Germany (5):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hamburg
- Novartis Investigative Site, Kopavogur, Iceland
- Novartis Investigative Site, London, United Kingdom

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=164

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 82 patients, male and female of non-childbearing potential aged 18-75 years, with Actinic Keratosis (AK) on the face or balding scalp were enrolled in the study.
Period: Overall Study
Arm/Group | LFX453 0.1% NMC | LFX453 0.15% LCC | Vehicle to NMC | Vehicle to LCC | Aldara
Started | 20 | 20 | 11 | 10 | 21
Completed | 18 | 20 | 10 | 9 | 18
Not Completed | 2 | 0 | 1 | 1 | 3
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 2
Not completed — Subject/guardian decision | 1 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LFX453 0.1% NMC | LFX453 0.15% LCC | Vehicle to NMC | Vehicle to LCC | Aldara | Total
Number analyzed (Participants) | 20 | 20 | 11 | 10 | 21 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (5.23) | 68.6 (6.25) | 68.3 (6.66) | 70.2 (4.32) | 68.6 (5.61) | 68.5 (5.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 0 | 2 | 0 | 9
  Male | 15 | 18 | 11 | 8 | 21 | 73

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events (AE)/Serious Adverse Events (SAE) as a Measure of Safety and Tolerability up to 20 Weeks
Description: Number of participants with at least one AE/SAE in the category up to 20 weeks
Time Frame: 20 weeks
Population: The safety analysis set included all patients that received any study drug. For Safety & Tolerability only the 2 vehicles have separate analysis.
Measure: Number; unit: participants
Arm/Group | LFX453 0.1% NMC | LFX453 0.15% LCC | Vehicle to NMC | Vehicle to LCC | Aldara
Number analyzed (Participants) | 20 | 20 | 11 | 10 | 21
participants
  Adverse Events (AEs) | 10 | 15 | 9 | 8 | 18
  Serious Adverse Events (SAEs) | 1 | 1 | 1 | 1 | 1

2. Primary Outcome: Number of Participants That Had Complete Clearance of Actinic Keratosis (AK) at 8 Weeks After the End of Treatment (Week 20) for LFX453 Compared to Vehicle Groups Combined
Description: Complete clearance of Actinic keratosis (AK), defined as the number of patients with a count of zero lesions in the treated area, evaluated 8 weeks after the end of treatment (Week 20) for LFX453 compared to vehicle groups combined
Time Frame: Week 20
Population: Pharmacodynamics (PD) analysis set included all patients with available PD data and no protocol deviations with relevant impact on PD data. For efficacy end points only there were combined analysis of the 2 vehicle groups. Vehicle groups were analyzed separately for safety and tolerability only.
Measure: Number; unit: participants
Groups:
- Combined Vehicle: Vehicle to nanomedicinal cream (NMC) and Vehicle to liquid crystal cream (LCC) Twice daily applications
Arm/Group | LFX453 0.1% NMC | LFX453 0.15% LCC | Combined Vehicle | Aldara
Number analyzed (Participants) | 20 | 20 | 21 | 21
participants | 1 | 1 | 1 | 13
Statistical Analysis 1: Comparison: LFX453 0.1% NMC vs Combined Vehicle; Test type: Non-Inferiority or Equivalence — p value is provided; p = 0.515, Posterior mean; Mean Difference (Net) = 0.00, 90% CI 2-sided [-0.12 to 0.12], Standard Deviation 0.07
Statistical Analysis 2: Comparison: LFX453 0.15% LCC vs Combined Vehicle; Test type: Non-Inferiority or Equivalence — p value is provided; p = 0.517, posterior mean; Mean Difference (Net) = 0.00, 90% CI 2-sided [-0.12 to 0.13], Standard Deviation 0.07

3. Secondary Outcome: Number of Participants That Had Complete Clearance of Actinic Keratosis (AK) at Week 8 and Week 16 for LFX453 Compared to Vehicle Groups Combined
Description: Complete clearance of Actinic keratosis (AK), defined as the number of patients with a count of zero lesions in the treated area, evaluated at week 8 and Week 16 for LFX453 compared to vehicle groups combined
Time Frame: week 8, week 16
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | LFX453 0.1% NMC | LFX453 0.15% LCC | Combined Vehicle | Aldara
Number analyzed (Participants) | 20 | 20 | 21 | 21
participants
  Week 8 | 0 | 0 | 1 | 3
  Week 16 | 1 | 1 | 1 | 9

4. Secondary Outcome: Number of Participants That Had Partial Clearance of Actinic Keratosis (AK) at 8 Weeks After the End of Treatment (Week 20) for LFX453 Compared to Vehicle Groups Combined
Description: Partial clearance of Actinic keratosis (AK), the defined as number of patients with at least 75% reduction in the number of AK lesion count compared to baseline, evaluated at 8 weeks after the end of treatment (Week 20 = EOS visit) for LFX453 compared to vehicle groups combined
Time Frame: Week 20
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | LFX453 0.1% NMC | LFX453 0.15% LCC | Combined Vehicle | Aldara
Number analyzed (Participants) | 20 | 20 | 21 | 21
participants | 1 | 2 | 2 | 16

5. Secondary Outcome: Number of Participants That Partial Clearance of Actinic Keratosis (AK) at at Week 8 and Week 16 for LFX453 Compared to Vehicle Groups Combined
Description: Partial clearance of Actinic keratosis (AK), the defined as number of patients with at least 75% reduction in the number of AK lesion count compared to baseline, evaluated at week 8 and Week 16 for LFX453 compared to vehicle groups combined
Time Frame: week 8, week 16
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | LFX453 0.1% NMC | LFX453 0.15% LCC | Combined Vehicle | Aldara
Number analyzed (Participants) | 20 | 20 | 21 | 21
participants
  Week 8 | 1 | 0 | 3 | 7
  Week 16 | 3 | 4 | 3 | 15

6. Primary Outcome: Reduction Rate (Percent) of Actinic Keratosis (AK) Lesion Count at 8 Weeks After the End of Treatment (Week 20) for LFX453 Compared to Vehicle Groups Combined
Description: Reduction rate (percent) of Actinic keratosis (AK) lesion count at 8 weeks after the end of treatment (Week 20) for LFX453 compared to vehicle groups combined
Time Frame: Baseline, Week 20
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | LFX453 0.1% NMC | LFX453 0.15% LCC | Combined Vehicle | Aldara
Number analyzed (Participants) | 20 | 20 | 21 | 21
percent change | 33.2 (31.19) | 34.5 (33.20) | 34.3 (33.31) | 86.7 (23.53)

7. Secondary Outcome: Reduction Rate (Percent) of Actinic Keratosis (AK) Lesion Count at Week 8 for LFX453 Compared to Vehicle Groups Combined
Description: Reduction rate (percent) of Actinic keratosis (AK) lesion count at Week 8 for LFX453 compared to vehicle groups combined
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | LFX453 0.1% NMC | LFX453 0.15% LCC | Combined Vehicle | Aldara
Number analyzed (Participants) | 20 | 20 | 21 | 21
percent change | 21.9 (36.18) | 21.9 (28.91) | 32.3 (33.55) | 55.8 (36.54)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | LFX453 0.1% NMC | LFX453 0.15% LCC | Vehicle to NMC | Vehicle to LCC | Aldara
Serious Adverse Events (participants affected / at risk) | 1/20 | 1/20 | 1/11 | 1/10 | 1/21
Other Adverse Events (participants affected / at risk) | 10/20 | 14/20 | 9/11 | 8/10 | 17/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LFX453 0.1% NMC (N=20) | LFX453 0.15% LCC (N=20) | Vehicle to NMC (N=11) | Vehicle to LCC (N=10) | Aldara (N=21)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
ABDOMINAL HERNIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
CEREBRAL INFARCTION (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
DEPRESSION (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LFX453 0.1% NMC (N=20) | LFX453 0.15% LCC (N=20) | Vehicle to NMC (N=11) | Vehicle to LCC (N=10) | Aldara (N=21)
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
INCREASED TENDENCY TO BRUISE (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
VESTIBULAR DISORDER (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
BLEPHARITIS (Eye disorders) | 0 | 1 | 0 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
APHTHOUS ULCER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
APICAL GRANULOMA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 3 | 0 | 1 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
TOOTHACHE (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
APPLICATION SITE COLDNESS (General disorders) | 1 | 0 | 0 | 0 | 0
APPLICATION SITE ERYTHEMA (General disorders) | 0 | 0 | 0 | 0 | 5
APPLICATION SITE PRURITUS (General disorders) | 0 | 0 | 0 | 1 | 2
APPLICATION SITE SCAB (General disorders) | 0 | 0 | 0 | 0 | 2
CHILLS (General disorders) | 0 | 0 | 1 | 0 | 1
FATIGUE (General disorders) | 0 | 0 | 1 | 0 | 2
HYPOTHERMIA (General disorders) | 0 | 0 | 0 | 1 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 1 | 0 | 0 | 0 | 3
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 0 | 0 | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
BRONCHITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0
CYSTITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
EYE INFECTION (Infections and infestations) | 1 | 1 | 0 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1
INFLUENZA (Infections and infestations) | 1 | 0 | 0 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 1 | 5 | 3 | 1 | 1
ORAL HERPES (Infections and infestations) | 0 | 1 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 0 | 1
RELAPSING FEVER (Infections and infestations) | 0 | 0 | 0 | 0 | 1
SINUSITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0
TINEA PEDIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
CORNEAL ABRASION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
EYELID INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
HEAD INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 1
LACERATION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
MUSCLE RUPTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
PERIORBITAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
ANTIPSYCHOTIC DRUG LEVEL INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0
BLOOD CREATININE INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0 | 0 | 1
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 | 0 | 0 | 0 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
MYOSCLEROSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0
PERIARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
SEBORRHOEIC KERATOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
AUTONOMIC NERVOUS SYSTEM IMBALANCE (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
BURNING SENSATION (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
DIZZINESS (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
HEADACHE (Nervous system disorders) | 0 | 0 | 2 | 0 | 1
POLYNEUROPATHY (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
POOR QUALITY SLEEP (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
SCIATICA (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
AGITATION (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
BURNOUT SYNDROME (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
RENAL CYST (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
BLISTER (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
ECZEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
HAEMATOMA (Vascular disorders) | 0 | 1 | 0 | 1 | 1
HYPERTENSION (Vascular disorders) | 0 | 1 | 1 | 0 | 0
THROMBOSIS (Vascular disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.